CLINICAL TRIAL: NCT07252947
Title: Stress and Anxiety Effects on Valuation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 25-01195
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Reward Value Level

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Aim 1: Socially Evaluated Cold Pressor Task (SECPT) (Experimental): Participants will be randomly assigned to complete the Socially Evaluated Cold Pressor Task (SECPT). Cortisol samples will be collected throughout the study session. All participants will then complete a Food Value Task, during which they will view a series of reward stimuli (snack foods) over alternating task blocks.
  Interventions: Behavioral: Socially Evaluated Cold Pressor Task (SECPT)
- Aim 1: Non-Stressful Control Task (Active Comparator): Participants will be randomly assigned to complete a non-stressful control task. Cortisol samples will be collected throughout the study session. All participants will then complete a Food Value Task, during which they will view a series of reward stimuli (snack foods) over alternating task blocks.
  Interventions: Behavioral: Non-Stressful Control Task
- Aim 2: Socially Evaluated Cold Pressor Task (SECPT) (Experimental): Participants will be randomly assigned to complete the SECPT. Cortisol samples will be collected throughout the study session. Participants will then complete the Image Value Task, during which they will view a series of positive, negative or neutral images over alternating task blocks.
  Interventions: Behavioral: Socially Evaluated Cold Pressor Task (SECPT)
- Aim 2: Non-Stressful Control Task (Active Comparator): Participants will be randomly assigned to complete a non-stressful control task. Cortisol samples will be collected throughout the study session. Participants will then complete the Image Value Task, during which they will view a series of positive, negative or neutral images over alternating task blocks.
  Interventions: Behavioral: Non-Stressful Control Task
- Aim 3: Socially Evaluated Cold Pressor Task (SECPT) (Experimental): Participants will first complete demographic and self-report measures, followed by random assignment to complete the SECPT. Cortisol samples will be collected throughout the study session to measure neuroendocrine response to the stress/control task. Participants will then complete the Affective Prediction Error Task.
  Interventions: Behavioral: Socially Evaluated Cold Pressor Task (SECPT)
- Aim 3: Non-Stressful Control Task (Active Comparator): Participants will be randomly assigned to complete a non-stressful control task. Cortisol samples will be collected throughout the study session. Participants will then complete the Affective Prediction Task.
  Interventions: Behavioral: Non-Stressful Control Task
- Aim 4: Behavioral Task (No Intervention): Participants with a diagnosis of generalized anxiety disorder (GAD) will complete a two-session behavioral task examining how clinical anxiety affects value and affective predictions.

INTERVENTIONS:
Behavioral: Socially Evaluated Cold Pressor Task (SECPT) — The SECPT is a validated laboratory stressor that combines physiological stress with social evaluative components; it is widely used to elicit acute stress responses in controlled settings. Participants are asked to submerge their nondominant hand into an ice-cold water (0-4°C) for 3 minutes, while videotaped and observed by one neutral-faced experimenter.
  Arms: Aim 1: Socially Evaluated Cold Pressor Task (SECPT); Aim 2: Socially Evaluated Cold Pressor Task (SECPT); Aim 3: Socially Evaluated Cold Pressor Task (SECPT)
Behavioral: Non-Stressful Control Task — Participants assigned to the warm water control condition will perform a non-evaluative task with warm water.
  Arms: Aim 1: Non-Stressful Control Task; Aim 2: Non-Stressful Control Task; Aim 3: Non-Stressful Control Task

SUMMARY:
The purpose of this study is to understand how stress, anxiety, and negative affect change learning and decision-making processes. The primary objective is to assess two forms of decision-making-reward adaptation and emotion prediction errors-differ as a function of stress and anxiety. The secondary objectives are to assess how individual differences measured in our studies relate to these decision variables.

ELIGIBILITY:
Inclusion Criteria:

Aims 1-3: To be eligible for participation in this study, an individual must meet all of the following criteria:

* 18-65 years of age
* Able to speak, read, and write fluently in English
* Be willing and able to follow study procedures and provide informed consent.

Aim 4: To be eligible for participation in this study, an individual must meet all of the following criteria:

* 18-65 years of age
* Diagnosis of GAD
* Able to speak, read, and write fluently in English
* Be willing and able to follow study procedures and provide informed consent.

Exclusion Criteria:

Aims 1-3: Individuals will be excluded from participation if any of the following criteria are met:

* History of or medication for neurologic or psychiatric disease
* High-blood pressure or heart condition
* Diabetes, food allergies, metabolic disorders or history of eating disorder
* Use of corticosteroids or beta-blockers
* Pregnancy

Aim 4: Individuals will be excluded from participation if any of the following criteria are met:

* High-blood pressure or heart condition
* Diabetes, food allergies, metabolic disorders or history of eating disorder
* Use of corticosteroids or beta-blockers
* Lifetime history of bipolar disorder or any psychotic disorder; substance use disorder in past 3 months; eating disorder in past 6 months; current major depressive disorder (past is allowed)
* Active suicidal ideation with plan and intent (indicated by score >=4 on the Columbia Suicide Severity Scale)
* Not on stable dose of psychiatric medication for at least 4 weeks prior to study participation
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2028-11-07 (Estimated); Study Completion 2028-11-07 (Estimated)

PRIMARY OUTCOMES:
Subjective Value Assigned to Food Stimuli | Study Visit (Day 1 - Approx. 2 Hours)
  Measured as participants' willingness-to-pay ($) for snack foods across the behavioral task. (Aims 1 and 4).
Valence Rating Score of OASIS Images | Study Visit (Day 1 - Approx. 2 Hours)
  Valence is rated on a scale from 0 (very negative) to 6 (very positive). (Aims 2 and 4)
Pleasantness Rating Score of OASIS Images | Study Visit (Day 1 - Approx. 2 Hours)
  Pleasantness is rated on a scale from 0 (very unpleasant) to 6 (very pleasant). (Aims 2 and 4)
Intensity Rating Score of OASIS Images | Study Visit (Day 1 - Approx. 2 Hours)
  Intensity is rated on a scale from 0 (very low) to 6 (very high). (Aims 2 and 4)
Emotion Predictions - Valence | Study Visit (Day 1 - Approx. 2 Hours)
  Difference in valence ratings before and after trial outcomes. (Aims 3 and 4)
Emotion Predictions - Pleasantness | Study Visit (Day 1 - Approx. 2 Hours)
  Difference in pleasantness ratings before and after trial outcomes. (Aims 3 and 4)

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) Score | Study Visit (Day 1 - Approx. 2 Hours)
  The PSS is a 10-item assessment of stressful feelings and thoughts over the past month; each item is rated on a 5-point Likert scale ranging from 0 (never) to 4 (fairly often). The total score is the sum of responses and ranges from 0-20. Higher scores indicate greater levels of perceived stress. (Aims 3 and 4)
Holmes-RaHe Life Stress Inventory Score | Study Visit (Day 1 - Approx. 2 Hours)
  Measurement of lifetime stress; comprises 43 items, each item represents a stressful event that may have occurred over the course of the participant's lifetime. The total score is the total number of stressful events that have occured; the total score ranges from 0-43; higher scores indicate greater lifetime stress. (Aims 3 and 4)
Multidimensional Assessment of Interoceptive Awareness (MAIA-2) Score | Study Visit (Day 1 - Approx. 2 Hours)
  The MAIA-2 is a 37-item assessment of interoceptive awareness. Each item is rated on a 6-point Likert scale from 0 (never) to 5 (always); the total score is the average of responses and ranges from 0 to 5; higher scores indicate greater equates to more awareness of bodily sensation.

CONTACTS AND LOCATIONS:
Overall Officials: Candace Raio, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data collected in this study will be used for upcoming grant submissions and not publication. We do not intend to share unpublished pilot data that goes into our grant proposals. The data collected in this study are used to acquire funding for a fully powered version of this pilot study.